CLINICAL TRIAL: NCT03275259
Title: Effect of Extracorporeal Shock Wave Therapy in the Treatment of Gynoid Lipodystrophy and Localized Fat
Brief Title: Shock Waves for Treatment of Gynoid Lipodystrophy and Localized Fat
Acronym: ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indústria Brasileira Equipamentos Médicos - IBRAMED (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ibramed -SW
Record Dates: First submitted 2017-07-21; First posted 2017-09-07 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Lipodystrophy; Cellulitis; Adiposity
Keywords: Shock wave; Gynoid lipodystrophy; Cellulits
MeSH Terms: conditions — Lipodystrophy; Cellulitis; Obesity

STUDY DESIGN:
Masking Description: The participants and evaluator are blinded. They will not be informed about the parameters applied in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracorporeal shock waves (Experimental): Composed of 30 female patients with glandular lipodystrophy in the buttocks and posterior thigh and fat located in abdomen and flanks that received the treatment of extracorporeal shock waves with energy between 100 and 180mJ, frequency of 15Hz and 6000 shots in abdomen, glutes and thigh Back and flanks 3000 shots with radial applicator and 15mm tip. The treatment is performed twice a week for 1 hour and 30 minutes each session.
  Interventions: Device: THORK Shock Wave® (Extracorporeal shock waves)

INTERVENTIONS:
Device: THORK Shock Wave® (Extracorporeal shock waves) — Treatment with extracorporeal shock waves: energy between 100 and 180mJ, frequency of 15Hz and 6000 shots in abdomen, glutes and thigh Back and flanks 3000 shots with radial applicator and 15mm tip. The treatment is performed twice a week for 1 hour and 30 minutes each session.

SUMMARY:
PURPOSE: To evaluate the efficacy of shock waves extracorporea in improving body contour,decrease fat localized and appearance of gynoid lipodystrophy.

SUBJECTS AND METHODS: A prospective and comparative longitudinal clinical study will be performed in 30 women with localized fat and gynoid lipodystrophy. Patients will be submitted data collection and assessments and before and after treatment.

HYPOTHESES: It is expected that the patients will present improvement in the body contour, decrease fat localized and in the picture of the gynoid lipodystrophy after of the therapies.

STATISTICAL ANALYSIS: A descriptive analysis will be done before and after vibration-oscillatory therapy, with frequency tables for categorical and descriptive variables (mean, standard deviation, median, minimum and maximum values) for continuous or numerical variables. In order to compare the main variables between the groups and the collection times, the analysis of variance (ANOVA) for repeated measurements will be used. Tukey's test will be used to compare groups. The level of significance adopted for the statistical tests will be 5% or p <0.05.

DETAILED DESCRIPTION:
After signing the informed consent, the participants will be evaluated by two physiotherapists where the data collected will be personal data, anthropometrics and complementary diagnostic tests, such as: ultrasound diagnosis to evaluate the thickness of the adipose tissue and Cutomiter analysis of the Viscoelasticity of skin. They then started treatment with another physiotherapist who will perform the following study protocol: placing a light layer of neutral gel on the treatment area, applying extracorporeal shock waves with the stainless steel tip with 180mJ of energy totaling 4 thousand shots , in abdomens, buttocks and posterior thigh and 2 thousand shots in flanks, then performs the change of the tip to the plastic and performs 2 thousand shots in the regions of abdomens, buttocks, posterior thigh emil shots in the region of flanks. The protocol will be performed twice a week for 1 and 20 hours each, totaling 10 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years of age up to premenopausal age (50 years of age).
* With body mass index considered eutrophic and / or overweight.
* Patients with lipodystrophy and localized abdominal fat.
* non smokers.
* Who agree to participate and sign the informed consent form.

Exclusion Criteria:

* Male gender.
* Possible.
* Haemophilia carriers and hemorrhagic disorders.
* Carriers diabetes mellitus.
* Women in menopause.
* Performed aesthetic treatment in the gluteal, thigh and abdominal regions in the last 1 months.
* Patients with skin lesions, such as dermatitis and dermatoses.
* Patients with acute deep vein thrombosis (DVT).
* About or close to cancerous lesions.
* Patients with cardiac pacemaker or other implanted electronic device.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Anthropometric evaluation | Ten minutes
  BMI (kg / height m2)
Anthropometric evaluation | Ten Minutes
  Perimeter in the region to be treated in centimeters.
Evaluation of the degree of cellulite | Ten minutes
  Assessment of Gland Lipodystrophy: Cellulite Severity Scale (CSS). Photographic study.
Assessment of adipose tissue thickness | Twenty minutes
  Assessment of the thickness of the dermis or hypodermis (Ultrasound diagnosis)
Assessment of skin elasticity | Twenty minutes
  Evaluation of skin elasticity (Cutometer® MPA580)

CONTACTS AND LOCATIONS:
Overall Officials: Débora O Modena, M.S, Principal Investigator — Ibramed - Industria Brasileira de Equipamentos Médicos
Locations (1):
- Ibramed - Indústria Brasileira de Equipamentos Médicos, Amparo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The data collected and the results of this study will be shared through scientific papers after the end of the study.

REFERENCES:
- [Background] Knobloch K, Joest B, Kramer R, Vogt PM. Cellulite and focused extracorporeal shockwave therapy for non-invasive body contouring: a randomized trial. Dermatol Ther (Heidelb). 2013 Dec;3(2):143-55. doi: 10.1007/s13555-013-0039-5. Epub 2013 Dec 3. PMID 24297647
- [Background] Adatto M, Adatto-Neilson R, Servant JJ, Vester J, Novak P, Krotz A. Controlled, randomized study evaluating the effects of treating cellulite with AWT/EPAT. J Cosmet Laser Ther. 2010 Aug;12(4):176-82. doi: 10.3109/14764172.2010.500392. PMID 20590369
- [Background] Kuhn C, Angehrn F, Sonnabend O, Voss A. Impact of extracorporeal shock waves on the human skin with cellulite: a case study of an unique instance. Clin Interv Aging. 2008;3(1):201-10. doi: 10.2147/cia.s2334. PMID 18488890
- [Background] Ferraro GA, De Francesco F, Cataldo C, Rossano F, Nicoletti G, D'Andrea F. Synergistic effects of cryolipolysis and shock waves for noninvasive body contouring. Aesthetic Plast Surg. 2012 Jun;36(3):666-79. doi: 10.1007/s00266-011-9832-7. Epub 2011 Nov 1. PMID 22042359
- [Background] Russe-Wilflingseder K, Russe E, Vester JC, Haller G, Novak P, Krotz A. Placebo controlled, prospectively randomized, double-blinded study for the investigation of the effectiveness and safety of the acoustic wave therapy (AWT((R))) for cellulite treatment. J Cosmet Laser Ther. 2013 Jun;15(3):155-62. doi: 10.3109/14764172.2012.759235. Epub 2013 May 21. PMID 23688206
- [Background] Siems W, Grune T, Voss P, Brenke R. Anti-fibrosclerotic effects of shock wave therapy in lipedema and cellulite. Biofactors. 2005;24(1-4):275-82. doi: 10.1002/biof.5520240132. PMID 16403988
- [Background] Schlaudraff KU, Kiessling MC, Csaszar NB, Schmitz C. Predictability of the individual clinical outcome of extracorporeal shock wave therapy for cellulite. Clin Cosmet Investig Dermatol. 2014 May 23;7:171-83. doi: 10.2147/CCID.S59851. eCollection 2014. PMID 24920933
- [Background] Christ C, Brenke R, Sattler G, Siems W, Novak P, Daser A. Improvement in skin elasticity in the treatment of cellulite and connective tissue weakness by means of extracorporeal pulse activation therapy. Aesthet Surg J. 2008 Sep-Oct;28(5):538-44. doi: 10.1016/j.asj.2008.07.011. PMID 19083577
- [Background] Nassar AH, Dorizas AS, Shafai A, Sadick NS. A randomized, controlled clinical study to investigate the safety and efficacy of acoustic wave therapy in body contouring. Dermatol Surg. 2015 Mar;41(3):366-70. doi: 10.1097/DSS.0000000000000290. PMID 25742559
- [Background] Milani GB, Natal Filho A, Amado Joao SM. Correlation between lumbar lordosis angle and degree of gynoid lipodystrophy (cellulite) in asymptomatic women. Clinics (Sao Paulo). 2008 Aug;63(4):503-8. doi: 10.1590/s1807-59322008000400015. PMID 18719762
- [Background] Pianez LR, Custodio FS, Guidi RM, de Freitas JN, Sant'Ana E. Effectiveness of carboxytherapy in the treatment of cellulite in healthy women: a pilot study. Clin Cosmet Investig Dermatol. 2016 Aug 22;9:183-90. doi: 10.2147/CCID.S102503. eCollection 2016. PMID 27578994
- [Background] Angehrn F, Kuhn C, Voss A. Can cellulite be treated with low-energy extracorporeal shock wave therapy? Clin Interv Aging. 2007;2(4):623-30. doi: 10.2147/cia.s1721. PMID 18225463
- [Derived] Modena DAO, Nogueira da Silva C, Delinocente TCP, Bianca de Araujo T, de Carvalho TM, Grecco C, Moreira RG, Campos G, de Souza JR, Michelini Guidi R. Effectiveness of the Electromagnetic Shock Wave Therapy in the Treatment of Cellulite. Dermatol Res Pract. 2019 Jun 20;2019:8246815. doi: 10.1155/2019/8246815. eCollection 2019. PMID 31320894